CLINICAL TRIAL: NCT03624153
Title: The Effects of the EMG-driven Exoskeleton Hand Robotic Training Device on Upper Extremity Motor and Physiological Function, Daily Functions, Quality of Life and Self-efficacy in Brain Injury Patients
Brief Title: The Effects of Exoskeleton Robotic Training Device on Upper Extremity in Brain Injury Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 201701543B0
Record Dates: First submitted 2018-08-07; First posted 2018-08-09 (Actual); Last update posted 2021-05-17 (Actual); Status verified 2020-01

CONDITIONS: Chronic Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robotic-assisted intervention (Experimental): 70 minutes Robotic-assisted intervention.
  Interventions: Behavioral: Robotic-assisted intervention
- Conventional intervention (Active Comparator): 70 minutes conventional rehabilitation.
  Interventions: Behavioral: Conventional rehabilitation intervention

INTERVENTIONS:
Behavioral: Robotic-assisted intervention — Participants received the 12-session robot-assisted intervention 3 sessions a week for 4 consecutive weeks. Each session consisted of 20-minute continuous passive motion, 20-minute active motion practice, and 30-minute task-oriented practice.
  Arms: Robotic-assisted intervention
Behavioral: Conventional rehabilitation intervention — Participants received the 12-session conventional rehabilitation intervention 3 sessions a week for 4 consecutive weeks. The intervention consisted of warm up including range of motion exercise, and strengthening exercise followed by task-oriented training for activities of daily living.
  Arms: Conventional intervention

SUMMARY:
The purpose of this study is to examine the effects of the EMG-driven exoskeleton hand robotic training device on upper extremity motor and physiological function, daily functions, quality of life and self-efficacy in brain injury patients.

DETAILED DESCRIPTION:
The purpose of this study was to 1) examine the effects of EMG-driven robot-assisted intervention, and 2) examine whether the robot-assisted therapy is as effective as conventional intervention. The study was conducted using a randomized, two-period crossover design. Participants were randomly assigned to group 1 or group 2 using a computer-generated list. Participants in group 1 received 12 sessions of robot-assisted intervention first, followed by a one-month washout period, and then received 12 sessions of conventional intervention. Participants in group 2 received 12 sessions of conventional intervention first, followed by a one-month washout period, and then received 12 sessions of robot-assisted intervention. Outcome measures were performed before the intervention, after the first 12-session intervention, and after the second 12-session intervention.

ELIGIBILITY:
Inclusion Criteria:

1. unilateral stroke ≥ 3 months prior to study enrollment
2. Fugl-Meyer Assessment for Upper Extremity (FMA-UE) score <60
3. without excessive spasticity in any of the UE joint (modified Ashworth scale ≤3)
4. Mini Mental State Exam (MMSE) score > 24, indicating no serious cognitive impairment
5. between the ages of 20 and 75 years.

Exclusion criteria:

1. histories of other neurological diseases such as dementia and peripheral polyneuropathy
2. difficulties in following and understanding instructions such as global aphasia
3. enroll in other rehabilitation or drug studies simultaneously
4. receiving Botulinum toxin injections within 3 months.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2018-07-30 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Change scores of Fugl-Myer Assessment (FMA) | Baseline, after completing the first 12-session intervention sessions (around 4 weeks after baseline); after completing the second 12-session intervention sessions (around 12 weeks after baseline
  The UE-FMA subscale will be used to assess the sensorimotor impairment level of UE in patients after stroke. The UE-FMA contains 33 movements with a score range from 0 to 66. A higher UE-FMA score indicates less impairment of the paretic limb. The validity and reliability of FMA is good to excellent.
Change scores of Wolf Motor Function Test (WMFT) | Baseline, after completing the first 12-session intervention sessions (around 4 weeks after baseline); after completing the second 12-session intervention sessions (around 12 weeks after baseline
  The WMFT is a reliable method to evaluate the UE motor ability in patients after stroke. The WMFT contains 15 function-based tasks and 2 strength-based tasks. The time (WMFT-time) and the functional ability (WMFT-quality) for an individual to complete the tasks will be recorded. A shorter WMFT-time and a larger WMFT-quality score indicate a faster movement and better quality of movement, respectively.
Change scores of Motor Activity Log (MAL) | Baseline, after completing the first 12-session intervention sessions (around 4 weeks after baseline); after completing the second 12-session intervention sessions (around 12 weeks after baseline
  The MAL will be used to assess the amount of use (AOU) and quality of movement (QOM) of the paretic UE. The MAL is a semi-structured interview that tests object manipulation and gross motor activities of daily living. The psychometric properties of MAL have been well-established, and a higher MAL score indicates better movement quality.
Change scores of Action Research Arm Test (ARAT) | Baseline, after completing the first 12-session intervention sessions (around 4 weeks after baseline); after completing the second 12-session intervention sessions (around 12 weeks after baseline
  The Action Research Arm Test (ARAT) evaluates 19 tests of arm motor function, both distally and proximally. Each test is given an ordinal score of 0, 1, 2, or 3, with higher values indicating better arm motor status. The total ARAT score is the sum of the 19 tests, and thus the maximum score is 57.

SECONDARY OUTCOMES:
Change scores of Mini-Mental State Exam (MMSE) | Baseline, after completing the first 12-session intervention sessions (around 4 weeks after baseline); after completing the second 12-session intervention sessions (around 12 weeks after baseline
  The Mini-Mental State Examination (MMSE) is the most commonly administered psychometric screening assessment of cognitive functioning. The MMSE is used to screen patients for cognitive impairment, track changes in cognitive functioning over time, and often to assess the effects of therapeutic agents on cognitive function. The total score of MMSE ranged from 0 to 30. Higher values represent a better cognitive functioning.
Change scores of Jamar hand dynamometer | Baseline, after completing the first 12-session intervention sessions (around 4 weeks after baseline); after completing the second 12-session intervention sessions (around 12 weeks after baseline
  The Jamar hand dynamometer is the most widely cited in the literature and accepted as the gold standard by which other dynamometers are evaluated. Excellent concurrent validity of the Jamar hand dynamometer is reported. The Jamar hand dynamometer measure the grip-strength. The norm of healthy male aged 18 to 75 years is from 64.8 lb to 121.8 lb, while the norm of healthy female aged 18 to 75 years is from 41.5 lb to 78.7 lb. Higher value represent a greater grip-strength.
Change scores of stroke self-efficacy questionnaire (SSEQ) | Baseline, after completing the first 12-session intervention sessions (around 4 weeks after baseline); after completing the second 12-session intervention sessions (around 12 weeks after baseline
  the Stroke Self-Efficacy Questionnaire (SSEQ) , a questionnaire developed to measure the most relevant self-efficacy and self-management domains specific to the stroke population. It contains 13 items that are rated on a 0 - 10 scale, with higher scores indicating greater levels of self-efficacy. Questionnaire includes a range of relevant functional tasks such as walking, getting comfortable in bed, as well as some self-management tasks.
Change scores of Modified Ashworth Scale (MAS) | Baseline, after completing the first 12-session intervention sessions (around 4 weeks after baseline); after completing the second 12-session intervention sessions (around 12 weeks after baseline
  The MAS is a 6-point ordinal scale that measures muscle spasticity in patients with brain lesions. Higher score indicates higher muscle tone. Investigators will assess the MAS scores of UE muscles, including biceps, triceps, wrist flexors and extensors, and finger flexors and extensors. The validity and reliability of MAS for patients with stroke were established to be adequate to good.
Change scores of Active Range of Motion (AROM) | Baseline, after completing the first 12-session intervention sessions (around 4 weeks after baseline); after completing the second 12-session intervention sessions (around 12 weeks after baseline
  Patient performs the exercise to move the joint without any assistance to the muscles surrounding the joint.

CONTACTS AND LOCATIONS:
Overall Officials: Ching-Yi Wu, Principal Investigator — Chang Gung University
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan, Taiwan

REFERENCES:
- [Derived] Chen YW, Chiang WC, Chang CL, Lo SM, Wu CY. Comparative effects of EMG-driven robot-assisted therapy versus task-oriented training on motor and daily function in patients with stroke: a randomized cross-over trial. J Neuroeng Rehabil. 2022 Jan 16;19(1):6. doi: 10.1186/s12984-021-00961-w. PMID 35034664